CLINICAL TRIAL: NCT05727735
Title: The Feasibility of Assessing Economic Costs of the Signia Stapler Versus Vessel Sealer Extend Energy Device With SureForm Stapling in Robotic-Assisted Segmentectomy for Lung Cancer
Brief Title: Signia Stapler Versus Vessel Sealer Extend Energy Device With SureForm Stapling in Robotic-Assisted Segmentectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Wael Hanna, Division Head & Associate Professor, Division of Thoracic Surgery, McMaster University, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15910
Record Dates: First submitted 2023-01-13; First posted 2023-02-14 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer; Thoracic Cancer; Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Medtronic Signia Stapler (Active Comparator): Patients randomized to this arm will undergo RTS segmentectomy with the Medtronic Signia Stapler.
  Interventions: Device: Medtronic Signia Stapler
- Da Vinci Vessel Sealer Extend Energy Device with SureForm Stapling (Experimental): Patients randomized to this arm will undergo RTS segmentectomy with the Da Vinci Vessel Sealer Extend Energy Device with SureForm Stapling.
  Interventions: Drug: Da Vinci Vessel Sealer Extend Energy Device with SureForm Stapling

INTERVENTIONS:
Device: Medtronic Signia Stapler — The Signia Stapler is a powered stapler that can be used for tissue dissection and vessel sealing during surgery.
  Arms: Medtronic Signia Stapler
Drug: Da Vinci Vessel Sealer Extend Energy Device with SureForm Stapling — The Vessel Sealer Extend Energy Device is integrated with the da Vinci system and uses bipolar energy technology to facilitate tissue dissection and vessel sealing.
  Arms: Da Vinci Vessel Sealer Extend Energy Device with SureForm Stapling

SUMMARY:
Robotic-assisted thoracoscopic surgery (RTS) segmentectomy is safe and effective for patients with early-stage non-small cell lung cancer (NSCLC). In RTS-segmentectomy, dissection and sealing procedures are performed by either staplers or energy devices.

Staplers, the current standard of care, have been associated with higher operating costs compared to energy devices for open lobectomy, RTS lobectomy and minimally invasive segmentectomy. However, there is a lack of prospective research evaluating the costs of the two methods for lung dissection and vessel sealing in RTS-segmentectomy.

This prospective trial seeks to determine whether it is feasible to conduct a randomized controlled trial evaluating the costs of the Signia stapler versus Vessel Sealer Extend energy device in RTS-segmentectomy for NSCLC. If this trial is feasible, we will be able to conduct a full-scale trial to compare costs and health outcomes, providing an economic evaluation that will inform hospital decision makers and clinicians in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 120 years at time of consent
* Ability to speak and understand English
* Clinical stage I, II or IIIa NSCLC
* Candidate for RTS segmentectomy, as determined by the operating surgeon

Exclusion Criteria:

* Anticoagulation with inability to cease anticoagulant therapy prior to surgery
* Incurable coagulopathy
* Systemic vascular disease or vasculitis
* Not a candidate for RTS segmentectomy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety | Up to 3 weeks post-surgery
  No adverse impacts of the study procedures on participants
Recruitment | Up to 8 weeks after recruitment first opens
  Recruitment rate of at least 70%
Randomization | Baseline
  Ability to randomize patients to one of two groups
Data collection of stapler reload model | Up to 3 weeks post-surgery
  Ability to collect the type of stapler reloads used
Data collection of stapler quantities | Up to 3 weeks post-surgery
  Ability to collect the number of stapler reloads used
Data collection of energy sealing data | Up to 3 weeks post-surgery
  Ability to collect the sealing time in seconds
Data collection of energy device data | Up to 3 weeks post-surgery
  Ability to collect the generator setting of the energy device

SECONDARY OUTCOMES:
Adverse events (AEs) and complications | 3 weeks post-surgery
  Short-term clinical outcomes, as measured by postoperative AEs and complications, will be recorded during patient follow-ups.
Intraoperative costs of stapler or energy device use | Up to 3 weeks following hospital discharge
  Surgical device (stapler or energy) costs per surgery will be collected and evaluated in Canadian dollars.
Hospitalization costs based on length of hospital stay | From admission to discharge, up to 14 days
  Inpatient hospitalization costs per day following surgery will be collected in Canadian dollars.

CONTACTS AND LOCATIONS:
Overall Officials: Waël C Hanna, MMDCM MBA FRCSC, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No